CLINICAL TRIAL: NCT06519201
Title: Effectiveness and Safety of SpineCare Used in Conjunction With Spinal Realignment Therapy in the Treatment of Idiopathic Scoliosis: An Investigator-initiated, Randomized, Single-blind, Pilot Study
Brief Title: Effectiveness and Safety of SpineCare Used in Conjunction With Spinal Realignment Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REBOM CLINIC (Other)
Responsible Party: Principal Investigator, Sohyun Kim, Dr. SH Kim, REBOM CLINIC
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RBIRB
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis Idiopathic
Keywords: Scoliosis; spinal realignment therapy
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRT with SpineCare (Experimental): The Trial Group underwent Spinal realignment therapy with SpineCare
  Interventions: Device: SRT with SpineCare
- SRT without SpineCare (Active Comparator): The Control Group underwent Spinal realignment therapy without SpineCare
  Interventions: Device: SRT without SpineCare

INTERVENTIONS:
Device: SRT with SpineCare — Korean medicine doctors performed the treatment regimens.The TG underwent SRT with SpineCare. Treat-ment was administered for six consecutive weeks, with sessions held twice per week dur-ing the first four weeks and once per week during the final two weeks. No additional treatments (e.g., procedures or surgeries) were allowed during the six-week period. To an-alyze pain according to the number of treatment sessions, a counselor assessed patients using the NRS after each of the ten treatment sessions. To compare the differences in Cobb's angle between the groups, X-rays were performed after the first and tenth treatment sessions. Detailed records of adverse events were maintained before and after each treat-ment session.
  Arms: SRT with SpineCare
Device: SRT without SpineCare — Korean medicine doctors performed the treatment regimens. The CG underwent SRT without SpineCare. Treat-ment was administered for six consecutive weeks, with sessions held twice per week dur-ing the first four weeks and once per week during the final two weeks. No additional treatments (e.g., procedures or surgeries) were allowed during the six-week period. To an-alyze pain according to the number of treatment sessions, a counselor assessed patients using the NRS after each of the ten treatment sessions. To compare the differences in Cobb's angle between the groups, X-rays were performed after the first and tenth treatment sessions. Detailed records of adverse events were maintained before and after each treat-ment session.
  Arms: SRT without SpineCare

SUMMARY:
* The goal of this study is to evaluate the safety and effectiveness of traction treatment using SpineCare Device.
* Research period: May 1, 2023 - November 30, 2023 (7 months)
* Research subjects

  * Male/female between 19 and 70 years old
  * Scoliosis patients: Scoliosis patients whose Cobb's angle is less than 15°~39°
* Treatment method: Group that applied traction treatment using SpineCare (traction device) and group that applied traction treatment without using SpineCare (traction device)
* Treatment period: Treatment twice a week from the 1st to 3rd week from the start of treatment, treatment once a week from the 4th to 7th week, A total of 10 times (takes approximately 2 months)
* Treatment time: approximately 50 minutes

DETAILED DESCRIPTION:
1. Introduction Idiopathic scoliosis (IS) is a condition characterized by an abnormal lateral curvature and rotational deformity of the vertebral column, typically presenting as either an S- or C-shaped curve in the vertebral column. IS leads to musculoskeletal asymmetry, culminating in morphological and geometric changes in the torso. It can result in numerous is-sues such as changes in posture, sensory impairment, balance and gait problems, limitations in physical activity, pain, body image disturbances, and challenges in social communication . The treatment approach for IS depends on the severity of the curve measured by Cobb's angle: surgical intervention is considered for angles of 40º or greater, while non-surgical treatments are considered for angles under 40º. Non-surgical modalities include physical therapy, manipulative therapy, braces, and exercise therapy. Traditionally, braces are recommended for Cobb's angles of 20-40º. However, braces often lead to undesirable effects such as psychological stress, discomfort in daily activities, negative selfesteem, and impaired respiratory function , and their effectiveness remains controversial . Manipulative therapy aims to correct the alignment of spinal segments and optimize the mechanical interaction between the spine and torso to facilitate healing and restore spinal mobility. Therefore, manipulative therapy focusing on correcting the position of spinal segments and improving neuromuscular stabilization is needed to manage IS [9]. Such treatments include chiropractic therapy, Chuna manual therapy (CMT), and spinal realignment therapy (SRT).

   The difference among these three treatment modalities is the patient's posture during treatment. During chiropractic treatment or CMT, the patient lies in the supine or prone position. During SRT, the patient lies in the prone position, and the lower extremities are placed under traction against gravity using SpineCare. SpineCare (Korea, Dr. Bom, Co., Ltd.) is a modernized traction device inspired by Panseo (攀索), which was introduced in the section on external therapy techniques (正骨心法要旨) in "Yizong Jinjian," a medical treatise compiled by Wu Jia (吳假) and others during the Qing Dynasty. This contraption received medical device certification from the Korean Ministry of Food and Drug Safety in 2020 (License No. 20-5054). The SpineCare device is used by having the patient lying prone with knees bent at 90º and both ankles secured on ankle braces to pull them up-wards against gravity. This posture helps create space between spinal segments, allowing deformed spinal and skeletal structures to return to their normal positions. With-out SpineCare, spinal imbalance may not be adequately addressed and corrected. Administering corrective treatment without spinal segment spacing may actually decrease spacing, increase pressure between the discs and vertebrae, and exacerbate disc abnormalities. Furthermore, it may affect the adjacent muscles and ligaments, thereby increasing pain and restricting movement and function, which, in turn, could cause discomfort and limitations in performing the activities of daily living. Thus, ensuring adequate space be-tween spinal segments using SpineCare is crucial for restoring the normal positions of the spine and skeletal structures.

   However, research on the effectiveness of SRT using SpineCare is insufficient. There-fore, this study aimed to assess the effectiveness and safety of the application of SRT in conjunction with SpineCare in patients with IS. In this study, we will elaborate on the specific procedures involved in SRT with SpineCare for patients with IS and report the out-comes using NRS and Cobb's angle.
2. Materials and Methods 2.1. Study Design and Setting This investigator-initiated, randomized controlled, single-blind trial was approved by the Institutional Review Board (Date of approval: Rebom Clinic June 1, 2023). Written informed consent was obtained from all patients before trial commencement.

2.2. Participants Participants were enrolled from among the patients of Rebom Clinic from June 1 to November 30, 2023, by posting a recruitment announcement within the clinic. The inclusion criteria were age ranging from 19-70 years and spinal radiographs obtained in an upright position. Patients with a Cobb's angle of 15-39º on X-rays who consented to participate in the trial were included. The exclusion criteria were spine-related surgery in the past six months, diagnosis of osteoporosis, history of other non-surgical treatments, participation in another interventional clinical trial in the past month (including human studies), and plan to participate in another interventional study after starting this trial.

2.3. Randomization and Allocation Concealment The investigator responsible for data analysis prepared two envelopes marked with odd and even numbers. Participants chose an envelope in the order of arrival. To maintain a 1:1 ratio between the trial and control groups, participants were assigned to the remaining group once one group reached capacity. Participants who chose an odd number were assigned to the SpineCare based SRT group (trial group, TG), and those who chose an even number were assigned to the SRT group without SpineCare (control group, CG).

2.4. Outcomes 2.4.1. Primary Outcome Measure The primary outcome was the Numerical Rating Scale (NRS) score, which was used to quantify the subjective pain experienced by the patient over the past week . Patients selected a number that best reflected their pain intensity, where 0 indicates no pain and 10 represents extreme pain, with higher values indicating greater severity of pain. There is consensus that the NRS has greater validity and intensity compared to other instruments . The Pearson correlation coefficient (r = 0.93) indicating the correlation be-tween the NRS and Visual Analog Scale indicates robust validity and reliability.

2.4.2. Secondary Outcome Measures The secondary outcome measure was Cobb's angle, which is typically used to assess the severity of scoliosis. Cobb's angle is defined as the angle between a line parallel to the upper border of the upper vertebra and a line parallel to the lower border of the lowermost vertebra of the lateral curvature of the spine . The inter-rater and intrarater reliability coefficients for measuring Cobb's angle are 0.970 and 0.969, respectively.

2.4.3 Safety Adverse events were monitored through patient interviews before and after treatment. Participants were also instructed to notify the medical team by phone any time upon occurrence of an adverse event.

2.5. Interventions Korean medicine doctors performed the treatment regimens for both groups. The TG underwent SRT with SpineCare, while the CG underwent SRT without SpineCare. Treat-ment was administered for six consecutive weeks, with sessions held twice per week dur-ing the first four weeks and once per week during the final two weeks . No additional treatments (e.g., procedures or surgeries) were allowed during the six-week period. To analyze pain according to the number of treatment sessions, a counselor assessed patients using the NRS after each of the ten treatment sessions. To compare the differences in Cobb's angle between the groups, X-rays were performed after the first and tenth treatment sessions. Detailed records of adverse events were maintained before and after each treat-ment session.

2.5.1. Spinal Realignment Therapy SRT, an original spinal alignment technique developed by the Society of Spinal Conduction Exercise and Manipulation, functions as a diagnostic and manual therapeutic technique to promote balance and improve harmony in the human body. In this study, SRT was implemented in three steps.

Step 1 entailed the application of traction. With the patient lying on their side, the practitioner grasps the leg on top at the dorsum and heel and slowly pulls it. This motion slightly dislocates the femoral head from the hip joint, allowing it to realign to its normal position, thereby relieving deformities in the hip joint and tension in the surrounding muscles and soft tissues. Next, the patient lies prone with knees bent. The ankles are then secured with SpineCare's ankle braces, and the knees are lifted slightly against gravity. In this position, the practitioner uses their hands or feet to apply frictional force, pushing the sacrum towards the direction of the coccyx to correct the former's position.

Step 2 entails the application of pressure and thrust. This step treats pelvic imbalance while the patient is prone with the lower limbs lifted against gravity. The practitioner places their hands or feet on the patient's right and left iliac crests, sacroiliac joints, and sacrum, using their body weight to exert pressure. This process aims to correct any misa-lignment of the sacrum and sacroiliac joints as well as the imbalance of the left and right ilia.

Step 3 entails securing the intervertebral space. The practitioner addresses the im-balance in the thoracolumbar region, while the patient remains prone with the lower limbs lifted against gravity. The practitioner applies pressure sequentially to the patient's deformed sacral spinous processes, lumbar spinous processes, and thoracic spinous pro-cesses using their hands or feet. This technique aims to align the position of the sacrum, the space between L5-S1, and the space between the facet joints and spinous processes of the lumbar and thoracic segments to their normal positions.

2.5.2. SpineCare In the TG, patients lay prone on the SpineCare mattress. When patients bend their knees, the practitioner secures both ankles in SpineCare's ankle braces. Next, the legs are lifted against gravity to a height of 1-5 cm above the floor till a point that does not strain the patient's pelvis based on the physician's judgment. In this position, steps 1-3 of the SRT are performed . After treatment, the legs are lowered to the floor using SpineCare's ankle braces.

The CG underwent steps 1-3 while lying prone on a regular therapy mattress .

2.6. Statistical Analysis Statistical analyses were performed using SPSS 18.0 for Windows (SPSS Inc., Chicago, IL, USA). NRS scores after each treatment session were compared (sessions 1-10). Data between the TG and CG were compared using Wilcoxon's signed-rank test and the Mann-Whitney U test. The values of Cobb's angle at baseline (session 1) and after the tenth treatment session were compared. All data were presented as the mean ± standard devia-tion or number (%). p-values <.05 were deemed statistically significant. Odds ratios were computed for comparison between the TG and CG, including the main analysis, and re-sults were deemed significant when the 95% confidence interval (CI) did not include 1. Adverse events were presented as frequencies and percentages, and the chi-squared test or Fisher's exact test (Fisher's exact test is used when more than 25% of the cells have an ex-pected frequency of less than 5) was used to compare the groups as needed.

ELIGIBILITY:
Inclusion Criteria:

* 19-70 years
* Patients with a Cobb's angle of 15-39º on X-rays who consented to par-ticipate in the trial were included.

Exclusion Criteria:

* spine-related surgery in the past six months,
* diagnosis of osteoporosis,
* history of other non-surgical treatments,
* participation in another interventional clinical trial in the past month

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) score | A total of 10 sessions from the start date of treatment (takes approximately 2 months)
  Patients selected a number that best reflected their pain intensity, where 0 indicates no pain and 10 represents extreme pain, with higher values indicating greater severity of pain.

SECONDARY OUTCOMES:
Cobb's angle | A total of 10 sessions from the start date of treatment (takes approximately 2 months)
  Cobb's angle is defined as the angle between a line parallel to the upper border of the upper vertebra and a line parallel to the lower border of the lowermost vertebra of the lateral curvature of the spine.

CONTACTS AND LOCATIONS:
Locations (1):
- Rebom Clinic, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schreiber S, Parent EC, Moez EK, Hedden DM, Hill D, Moreau MJ, Lou E, Watkins EM, Southon SC. The effect of Schroth exercises added to the standard of care on the quality of life and muscle endurance in adolescents with idiopathic scoliosis-an assessor and statistician blinded randomized controlled trial: "SOSORT 2015 Award Winner". Scoliosis. 2015 Sep 18;10:24. doi: 10.1186/s13013-015-0048-5. eCollection 2015. PMID 26413145
- [Result] Yagci G, Ayhan C, Yakut Y. Effectiveness of basic body awareness therapy in adolescents with idiopathic scoliosis: A randomized controlled study1. J Back Musculoskelet Rehabil. 2018;31(4):693-701. doi: 10.3233/BMR-170868. PMID 29630516
- [Result] Le Berre M, Guyot MA, Agnani O, Bourdeauducq I, Versyp MC, Donze C, Thevenon A, Catanzariti JF. Clinical balance tests, proprioceptive system and adolescent idiopathic scoliosis. Eur Spine J. 2017 Jun;26(6):1638-1644. doi: 10.1007/s00586-016-4802-z. Epub 2016 Nov 14. PMID 27844226
- [Result] Negrini S, Grivas TB, Kotwicki T, Maruyama T, Rigo M, Weiss HR; Members of the Scientific society On Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT). Why do we treat adolescent idiopathic scoliosis? What we want to obtain and to avoid for our patients. SOSORT 2005 Consensus paper. Scoliosis. 2006 Apr 10;1:4. doi: 10.1186/1748-7161-1-4. PMID 16759352
- [Result] Durmala J, Blicharska I, Drosdzol-Cop A, Skrzypulec-Plinta V. The Level of Self-Esteem and Sexual Functioning in Women with Idiopathic Scoliosis: A Preliminary Study. Int J Environ Res Public Health. 2015 Aug 12;12(8):9444-53. doi: 10.3390/ijerph120809444. PMID 26274967
- [Result] Koumbourlis AC. Scoliosis and the respiratory system. Paediatr Respir Rev. 2006 Jun;7(2):152-60. doi: 10.1016/j.prrv.2006.04.009. Epub 2006 Jun 2. PMID 16765303
- [Result] Negrini S, Carabalona R. Social acceptability of treatments for adolescent idiopathic scoliosis: a cross-sectional study. Scoliosis. 2006 Aug 24;1:14. doi: 10.1186/1748-7161-1-14. PMID 16930488
- [Result] Kuru T, Yeldan I, Dereli EE, Ozdincler AR, Dikici F, Colak I. The efficacy of three-dimensional Schroth exercises in adolescent idiopathic scoliosis: a randomised controlled clinical trial. Clin Rehabil. 2016 Feb;30(2):181-90. doi: 10.1177/0269215515575745. Epub 2015 Mar 16. PMID 25780260
- [Result] Burger M, Coetzee W, du Plessis LZ, Geldenhuys L, Joubert F, Myburgh E, van Rooyen C, Vermeulen N. The effectiveness of Schroth exercises in adolescents with idiopathic scoliosis: A systematic review and meta-analysis. S Afr J Physiother. 2019 Jun 3;75(1):904. doi: 10.4102/sajp.v75i1.904. eCollection 2019. PMID 31206094
- [Result] Reilly JP, Gersten JW, Clinkingbeard JR. Effect of pelvic-femoral position on vertebral separation produced by lumbar traction. Phys Ther. 1979 Mar;59(3):282-6. doi: 10.1093/ptj/59.3.282. PMID 419172
- [Result] Mathews JA. Dynamic discography: a study of lumbar traction. Ann Phys Med. 1968 Aug;9(7):275-9. doi: 10.1093/rheumatology/9.7.275. No abstract available. PMID 5676680
- [Result] Hood LB, Chrisman D. Intermittent pelvic traction in the treatment of the ruptured intervertebral disk. Phys Ther. 1968 Jan;48(1):21-30. doi: 10.1093/ptj/48.1.21. No abstract available. PMID 5636246
- [Result] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Result] Turk DC, Rudy TE, Sorkin BA. Neglected topics in chronic pain treatment outcome studies: determination of success. Pain. 1993 Apr;53(1):3-16. doi: 10.1016/0304-3959(93)90049-U. PMID 8316386
- [Result] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Result] Gstoettner M, Sekyra K, Walochnik N, Winter P, Wachter R, Bach CM. Inter- and intraobserver reliability assessment of the Cobb angle: manual versus digital measurement tools. Eur Spine J. 2007 Oct;16(10):1587-92. doi: 10.1007/s00586-007-0401-3. Epub 2007 Jun 5. PMID 17549526
- [Result] Park SY, Hwang EH, Cho JH, Kim KW, Ha IH, Kim MR, Nam K, Lee MH, Lee JH, Kim N, Shin BC. Comparative Effectiveness of Chuna Manipulative Therapy for Non-Acute Lower Back Pain: A Multi-Center, Pragmatic, Randomized Controlled Trial. J Clin Med. 2020 Jan 5;9(1):144. doi: 10.3390/jcm9010144. PMID 31948083
- [Result] Stokes IA, Burwell RG, Dangerfield PH; IBSE. Biomechanical spinal growth modulation and progressive adolescent scoliosis--a test of the 'vicious cycle' pathogenetic hypothesis: summary of an electronic focus group debate of the IBSE. Scoliosis. 2006 Oct 18;1:16. doi: 10.1186/1748-7161-1-16. PMID 17049077
- [Result] Huh S, Eun LY, Kim NK, Jung JW, Choi JY, Kim HS. Cardiopulmonary function and scoliosis severity in idiopathic scoliosis children. Korean J Pediatr. 2015 Jun;58(6):218-23. doi: 10.3345/kjp.2015.58.6.218. Epub 2015 Jun 22. PMID 26213550
- [Result] Saraiva BMA, Araujo GS, Sperandio EF, Gotfryd AO, Dourado VZ, Vidotto MC. Impact of Scoliosis Severity on Functional Capacity in Patients With Adolescent Idiopathic Scoliosis. Pediatr Exerc Sci. 2018 May 1;30(2):243-250. doi: 10.1123/pes.2017-0080. Epub 2017 Nov 28. PMID 28872419
- [Result] Bruyneel AV, Chavet P, Ebermeyer E, Mesure S. Idiopathic scoliosis: relations between the Cobb angle and the dynamical strategies when sitting on a seesaw. Eur Spine J. 2011 Feb;20(2):247-53. doi: 10.1007/s00586-010-1574-8. Epub 2010 Sep 19. PMID 20853120
- [Result] Walker BF, French SD, Grant W, Green S. A Cochrane review of combined chiropractic interventions for low-back pain. Spine (Phila Pa 1976). 2011 Feb 1;36(3):230-42. doi: 10.1097/BRS.0b013e318202ac73. PMID 21248591
- [Result] Rubinstein SM, van Middelkoop M, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for chronic low-back pain. Cochrane Database Syst Rev. 2011 Feb 16;2011(2):CD008112. doi: 10.1002/14651858.CD008112.pub2. PMID 21328304